CLINICAL TRIAL: NCT03199209
Title: Tu Salud ¡Si Cuenta! (Your Health Matters!): Promoting Healthy Lifestyles in Latino Family Dyads
Brief Title: Your Health Matters! (Tu Salud ¡Si Cuenta!): Promoting Healthy Lifestyles in Latino Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0399; NCI-2019-02503 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0399 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Family Member; Health Status Unknown
Keywords: physical activity; healthy eating; behavioral intervention; community health worker; Hispanic/Latino
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (home visit, information about healthy lifestyles) (Experimental): Participants and their family member meet with a community health worker in their home over 90 minutes to learn about physical activity, healthy eating, and to set goals, once a month for 6 months. Participants also receive 2-5 text messages per week that contain health tips related to healthy lifestyles and information about local resources. Participants also attend a study visit with a research staff over 90-120 minutes at a community center, MD Anderson, or at home at baseline, 6 months, and 12 months.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Behavioral: Patient Visit; Other: Questionnaire Administration; Other: Text Message
- Group II (home visit, information about healthy homes) (Experimental): Participants and their family member meet with a community health worker in their home over 90 minutes to receive information on how to be safe and healthy at home and information about indoor air quality, home safety, CPR/first aid, how to prepare for emergencies, and keeping pests away, once a month for 6 months. Participants also receive 2-5 text messages per week that contain information about healthy homes and local resources. Participants also attend a study visit with a research staff over 90-120 minutes at a community center, MD Anderson, or at home at baseline, 6 months, and 12 months.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Behavioral: Patient Visit; Other: Questionnaire Administration; Other: Text Message

INTERVENTIONS:
Other: Behavioral, Psychological or Informational Intervention — Receive information about healthy lifestyles
  Arms: Group I (home visit, information about healthy lifestyles)
Other: Behavioral, Psychological or Informational Intervention — Receive information about healthy homes
  Arms: Group II (home visit, information about healthy homes)
Behavioral: Patient Visit — Attend study visit with research staff
  Other Names: Healthcare Visit; Patient Encounter; Subject Visit; visit
Other: Questionnaire Administration — Ancillary studies
Other: Text Message — Receive information about healthy lifestyles
  Other Names: Text; SMS Text Message; SMS Text
  Arms: Group I (home visit, information about healthy lifestyles)
Other: Text Message — Receive texts about healthy homes
  Other Names: Text; SMS Text Message; SMS Text
  Arms: Group II (home visit, information about healthy homes)

SUMMARY:
This trial studies how well a theoretically-based motivational behavior change program called Tu Salud Si Cuenta! works in promoting healthy lifestyles in Latino families. Tu Salud Si Cuenta! will deliver programs on healthy lifestyles and healthy homes to Hispanic/Latino families and may help to improve their health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of the Tu Salud, Si Cuenta! Familiar (TSSC-Family) intervention in facilitating positive changes in physical activity and nutrition among Latino adults not meeting physical activity or nutrition recommendations.

SECONDARY OBJECTIVES:

I. To test the effects of TSSC-Family on hypothesized intervention mechanisms (e.g., self-efficacy, stage of change, social support, social control), and the role of those mechanisms in mediating TSSC-Family effects of physical activity and nutrition outcomes.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants and their family member meet with a community health worker in their home over 90 minutes to learn about physical activity, healthy eating, and to set goals, once a month for 6 months. Participants also receive 2-5 text messages per week that contain health tips related to healthy lifestyles and information about local resources. Participants also attend a study visit with a research staff over 90-120 minutes at a community center, MD Anderson, or at home at baseline, 6 months, and 12 months.

GROUP II: Participants and their family member meet with a community health worker in their home over 90 minutes to receive information on how to be safe and healthy at home and information about indoor air quality, home safety, cardiopulmonary resuscitation (CPR)/first aid, how to prepare for emergencies, and keeping pests away, once a month for 6 months. Participants also receive 2-5 text messages per week that contain information about healthy homes and local resources. Participants also attend a study visit with a research staff over 90-120 minutes at a community center, MD Anderson, or at home at baseline, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Hispanic/Latino ethnicity.
* Speak English or Spanish.
* Physically able to engage in low-to-moderate physical activity (PA) as assessed by the PA Readiness Questionnaire (PAR-Q), or with medical clearance.
* Insufficient self-reported moderate-to-vigorous PA (< 150 minutes/week) or limited fruits and vegetable (FV) intake (defined as less than or equal to 4 cups of FV combined or < 1 cup of vegetables per day).
* Able to enroll with one eligible adult family member.
* Valid home address in the Houston neighborhoods of Gulfton, the East End/Magnolia, Northside, Pasadena or adjacent neighborhoods.
* Have a functioning cellular telephone and able and willing to send and receive text messages.
* Blood pressure reading less than 160/100 mmHg, or with medical clearance.

Exclusion Criteria:

* Pregnancy or considering pregnancy during the study period, self-reported.
* Currently participating in a program or research study to promote physical activity, healthy eating, or weight loss.
* Plans to move outside the greater Houston area during the study period.
* Past weight loss surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-06-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Physical Activity | 12 months
  Changes in physical activity determined by using univariable and multivariable mixed effect models.
Increase in Fruit and Vegetable (F/V) Consumption | 12 months
  Assuming 1.6 portions of F/V consumed per day in the control group, power calculations show that Poisson regression model with a 0.05 two-sided significance level has 80% power to detect a 22% or greater increase (rate ratio (RR) =1.22) in portions of F/V consumption for intervention group if we have total 522 participants (261 dyads) with Intra-cluster correlation coefficient (ICC) of 0.08.

CONTACTS AND LOCATIONS:
Overall Officials: Larkin Strong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org